CLINICAL TRIAL: NCT06862817
Title: Comparison Between the Effect of Aloe Vera and Benzydamine Hydrochloride Mouth Gel on Radiation-induced Oral Mucositis (Randomized Clinical Trial)
Brief Title: Comparison Between the Effect of Aloe Vera and Benzydamine Hydrochloride Mouth Gel on Prevention of Pain and Progression of Radiation-induced Oral Mucositis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Minia University (Other)
Collaborators: Faculty of Medicine, Minia University (Unknown)
Responsible Party: Principal Investigator, Arwa Abdelrady Osman, resident, Minia University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Aloevera & benzydmin on RIOM
Record Dates: First submitted 2025-02-16; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Radiation Indused Oral Mucositis
Keywords: RIOM; aloevera; benzydamine; bioadhesive; mucositis
MeSH Terms: conditions — Mucositis | interventions — Aloe vera gel; Benzydamine; Gels

STUDY DESIGN:
Intervention Model Description: The patients divided into three groups, randomly selected for treatment:
  Group A: 1. Aloe vera mouth gel will be applied to areas affected by oral mucositis.
  Group B: benzydamine hydrochloride mouth gel will be applied to areas affected by oral mucositis.
  Group C: placebo mouth gel will be applied to areas affected by oral mucositis Treatment was given written instructions to apply with 2 mg of the gel and not eat or drink for the subsequent 30 min, 3 times a day from the last second week of RT for the 7 th week.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- benzydamine hydrochloride mouth gel (Active Comparator): found that benzydamine mouth rinses and gels could prevent or reduce the severity of oral mucositis.
  Interventions: Drug: Benzydamine Hydrochloride 0.15% Oral gel
- aloe vera gel (Active Comparator)
  Interventions: Drug: Aloe vera gel
- bioadhesive gel (Placebo Comparator): . They incorporate biodegradable mucoadhesive polymers to enhance retention on active mucosal surfaces and regulate the release of the drug
  Interventions: Drug: Aloe vera gel; Drug: bioadhesive gel

INTERVENTIONS:
Drug: Aloe vera gel — Aloe vera mouthgel not only as a potent agent for prevention mucositis, but also as a prevention of candidiasis in patients undergoing radiotherapy of head and neck with its antifungal and immunomodulation properties
  Arms: aloe vera gel; bioadhesive gel
Drug: Benzydamine Hydrochloride 0.15% Oral gel — . Benzydamine's mechanisms of action are rooted in its anti-inflammatory, anesthetic, and analgesic properties. It has been shown to reduce the synthesis of TNF-α, IL-1β and prostaglandins while also acting as an antioxidant by scavenging reactive oxygen species (ROS) benzydamine inhibits leukocyte-endothelial interactions, thereby decreasing neutrophil degranulation, and helps mitigate histamine-induced vasodilation and vascular permeability.
  Arms: benzydamine hydrochloride mouth gel
Drug: bioadhesive gel — bioadhesive These polymers increase viscosity through a liquid-to-semi-solid phase transition, improving retention at the administration site and providing a sustained release profile ,Mucoadhesive Dosage Forms These dosage forms are typically employed to administer medications to epithelial surfaces, including the buccal cavity, sublingual area, oral cavity, eyes, nasal passages, vagina, and lungs
  Arms: bioadhesive gel

SUMMARY:
Oral mucositis, a painful inflammation and ulceration of the mucous membranes in the mouth, is commonly seen in patients undergoing chemotherapy or radiation therapy. Effective management of this condition is crucial to reduce pain, promote healing, and maintain oral function.

Benzydamine mouth gel is a non-steroidal anti-inflammatory drug (NSAID) with analgesic and anti-inflammatory properties, making it useful in treating oral mucositis. It works by blocking pain and reducing inflammation, helping to relieve symptoms like soreness and swelling. Studies suggest that benzydamine gel can decrease the severity of mucositis, ease discomfort, and improve patients' quality of life.

Aloe vera gel is well-known for its soothing, anti-inflammatory, and wound-healing properties. When applied to oral mucositis lesions, it promotes healing by providing hydration and forming a protective barrier over the affected tissue. Aloe vera's natural compounds, such as glycoproteins and polysaccharides, help in pain relief and accelerate tissue repair, making it a complementary option to reduce mucositis severity.

Together, benzydamine and aloe vera gels can be effective in managing oral mucositis. Benzydamine offers immediate pain relief and reduces inflammation, while aloe vera aids in longer-term healing and tissue regeneration. This combination approach has shown promise in enhancing comfort and accelerating recovery for patients with mucositis.

DETAILED DESCRIPTION:
Head and neck cancer (HNC) is a broad term, including epithelial malignancies that occur in the paranasal sinuses, nasal cavity, oral cavity, pharynx, and larynx. Almost all these malignancies are head and neck squamous cell carcinoma (HNSCC).

HNSCC is the sixth most common cancer worldwide, with 890,000 new cases and 450,000 deaths in 2018. The principal modalities of curative therapy for locally or locoregionally confined HNSCC are resection, radiation and systemic therapy. Treatment planning should aim for the most highly curative approach, while optimizing preservation of function

Head and neck cancers (HNC) are often treated with radiation therapy (RT), a technique that utilizes ionizing radiation and exerts therapeutic effect by semi-selectively damaging the genetic material of vulnerable malignant cells, either directly or through the production of free radicals, resulting in cell death.

Radiation-induced oral mucositis (RIOM) is one of the major ionizing radiation toxicities and normal tissue injuries that result from radiotherapy. RIOM is a normal tissue injury lasting between 7 and 98 days, which starts as an acute inflammation of oral mucosa, tongue, and pharynx after RT exposure.

Oral mucositis is defined as inflammation of oral mucosa resulting from cancer therapy typically manifesting as atrophy, swelling, erythema and ulceration. The condition may be exacerbated by local factors, such as trauma from teeth, or microbial colonization. The term stomatitis refers to any inflammatory condition of oral tissue, including mucosa, dentition/periapices, and periodontium. Stomatitis thus defines a broader range of pathoses of oral tissues, including mucositis.

Treatment interruption may be required in patients who develop severe OM as further radiotherapy may lead to permanent loss of the stem cells and morbidity to treatment. But it should be noted that interruption of treatment is at the cost of reduced local control and may be compromised survival. Hence, it is important to have a balance of these factors when thinking of interrupting the treatment. It is also important that treatment is restarted at the earliest so that there is minimum gap in the treatment.

Currently, there is no definite efficient therapy for mucositis or its pain Multiple studies have been performed to propose preventive and therapeutic management. implementing proper oral hygiene measure ,removal of local irritants, and frequent rinsing with combination therapies are the current main supportive measure to mollify the severity of oral mucositis and reduce its attributed risk.

Numerous adjunctive treatments for the prevention of chemotherapy and radiotherapy -induced mucositis are now being studied such as the administration of honey, zinc, selenium, topical vitamin E, and glutamine .

Lalla RV recommend the use of benzydamine oral rinse for prevention of radiation induced OM in HNC patients treated with moderate doses of radiation therapy.

Aloe vera (named Aloe barbadensis in Latin), contains polysaccharides, anthraquinone, lectin, superoxide dismutase (an antioxidant enzyme), glycoprotein, amino acids, vitamins C and E and minerals. revealed the anti inflammatory, analgesic, liver protection, antiproliferative, anticarcinogenic and antiaging properties .

ELIGIBILITY:
Inclusion Criteria:

1. patients diagnosed by head and neck cancer indicated for radiotheraby treatment
2. Adult age range from 20-55 male and female patients.
3. The patients had receiving a total external-beam RT dose of at least 50 Gy in standard fractions where the oral cavity had been exposed to RT.
4. The Karnovsky performance status was more than 70%.
5. - Must be able to diffuse gel on oral cavity

Exclusion Criteria:

1. Food allergy.
2. Hypersensitivity to benzydamine or typical nonsteroidal anti-inflammatory drugs (NSAIDs).
3. Patients who had an existing lesion in the oral cavity (e.g. active infection or ulcer) before staring RT, or those who were unwilling to participate.
4. immunedifictincy desease

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
to compere the effect of Aloe vera mouth gel versus benzydamine mouth gel In the Management of pain and progression of Toxicity grading of oral mucositis according to World Health Organization (WHO) and National Cancer Institute Common Toxicity Criteria | from begining of radiation theraby at baseline and for 6 week ,once every one week
  A complete oral examination will be performed within 24 hours of the first dose of study medication and at each visit. Oral areas at risk will be scored for the major signs of oral mucositis (i.e., erythema, pseudomembrane, and ulceration) -Grade 0: no sighns or symptoms
  * Grade 1(mild) Oral soreness, erythema of mucosa.
  * Grade 2 (moderate)Oral erythema, ulcers, Patchy pseudomembranous reaction (patches generally ≤1.5 cm in diameter and non-contiguous),but can eat or swallow.
  * Grade 3 (severe):Confluent pseudomembranous reaction (contiguous patches generally >1.5 cm in diameter) requiring intravenous hydration.
  * Grade 4(life threatening): Necrosis or deep ulceration; may include bleeding not induced by minor trauma or abrasion.

CONTACTS AND LOCATIONS:
Locations (1):
- Arwa Abdelrady, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daugelaite G, Uzkuraityte K, Jagelaviciene E, Filipauskas A. Prevention and Treatment of Chemotherapy and Radiotherapy Induced Oral Mucositis. Medicina (Kaunas). 2019 Jan 22;55(2):25. doi: 10.3390/medicina55020025. PMID 30678228
- See also: Benzydamine mechanisms of action reside in its anti-inflammatory, anaesthetic and analgesic nature. It has been demonstrated that it may act both by decreasing TNF-α, IL-1β and prostaglandin synthesis and as an antioxidant (ROS scavenger). — https://link.springer.com/article/10.1007/s00520-021-06048-5